CLINICAL TRIAL: NCT06376318
Title: Beyond the Syndromic Approach in Critical Care: Identifying Biomarker-driven Subphenotypes of Circulatory Shock
Brief Title: Shock and Acute Conditions OutcOmes Platform
Acronym: ShockCO-OP
Status: Active, not recruiting | Type: Observational
Sponsor: Saint-Louis Hospital, Paris, France (Other)
Collaborators: University of Helsinki (Other); University of Ottawa (Other); University of Leipzig (Other); University of Nancy (Other); McGill University (Other); Mayo Clinic (Other); University of Paris 5 - Rene Descartes (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Sabri SOUSSI, Assistant Professor, University of Toronto
Other Study IDs: 19-138
Record Dates: First submitted 2024-04-01; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Circulatory Shock; Sepsis; Cardiogenic Shock; Major Trauma; Surgical Shock
Keywords: shock; heterogeneity of treatment effect; biomarkers; machine learning
MeSH Terms: conditions — Shock; Sepsis; Shock, Cardiogenic; Shock, Surgical | interventions — Vasoconstrictor Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Inotrope — Vasopressors: Norepinephrine, vasopressin Inotropes: Epinephrine, Dobutamine, Milrinone
  Other Names: Vasopressor
Device: Mechanical circulatory support — Intra-aortic balloon pump Extracorporeal membrane oxygenation (ECMO)
Drug: anti-bodies — Anti-Dipeptidyl peptidase 3 (DPP3), Anti-Bioactive adrenomedullin (bio-ADM)

SUMMARY:
In-hospital mortality of patients admitted in the intensive care unit (ICU) for circulatory shock remains high (between 20 and 40%).

Currently, there are no markers that allow us to classify patients with circulatory shock at higher risk of early and late bad outcomes, or who may better respond to a specific intervention.

To understand the contribution of biological heterogeneity to circulatory shock independently from its etiology, the ShockCO-OP Research Program aims to use clustering approaches to re-analyze existing clinical and molecular data from several large European and North American prospective cohorts and clinical trials.

This will enable an improvement in risk prediction and a better patient selection in future clinical trials to assess a personalized therapy (i.e., prospective enrollment based on a biological/molecular signature).

DETAILED DESCRIPTION:
Traditionally, circulatory shock subgroups are defined according to hemodynamic profile (e.g., hypovolemic, distributive, cardiogenic) and etiology (e.g., trauma, infection, myocardial infarction among others) and are incorrectly considered as homogeneous clinical syndromes. Emerging translational evidence highlights the existing molecular heterogeneity in the circulatory shock syndrome. Such findings raise a major issue in assessing neutral clinical trial results in circulatory shock as a given intervention effect (e.g., fluid management, vasopressors/inotropes, mechanical circulatory support) may preferentially impact different subgroups (i.e., heterogeneity of treatment effect).

Accordingly, identifying distinct biological subphenotypes with different mechanistic signatures may provide new insights regarding the pathophysiology of circulatory shock. This may allow predictive enrichment (i.e., identifying those patients most likely to benefit from a particular therapy) and biomarker-driven or phenotype-driven patient selection in future clinical trials to assess a personalized therapy (i.e., prospective enrollment based on a biological signature).

The ShockCO-OP Research Program aims to use unsupervised model-based clustering (i.e., regardless of outcome) to reanalyze existing clinical and biological data in several European and North American prospective cohorts and clinical trials to identify distinct biomarker-driven subphenotypes in circulatory shock syndromes, their underlying molecular signatures (proteomics, transcriptomics), their association with outcome and their response to different interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with circulatory shock on admission (i.e., the reported main cause of admission is septic shock, cardiogenic shock or hypovolemic/hemorrhagic shock).
2. Patients who required vasopressors infusion and presented signs of tissue hypoperfusion (e.g., altered mental state (Glasgow coma scale≤ 14), oliguria (urine output of < 0.5 ml/kg/h for at least six hours) or a serum lactate level of ≥2 mmol/l) within the first 24 h after admission.

Exclusion Criteria:

1. Mechanical circulatory support on admission
2. Serious arrythmia (e.g., rapid atrial fibrillation or ventricular tachycardia/fibrillation) on admission
3. Deceased patients within the first 24 hours after admission.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with circulatory shock on admission independently from its etiology
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 28 days

SECONDARY OUTCOMES:
Mortality rate | 1 year
Renal replacement therapy use rate | 28 days
Mechanical circulatory support use rate | 28 days
Vasopressors and inotropes-free days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Claudia dos Santos, MD, PhD, Principal Investigator — Unity Health Toronto; Alexandre Mebazaa, MD, PhD, Study Chair — St Louis and Lariboisiere Hospitals
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Soussi S, Dos Santos C, Jentzer JC, Mebazaa A, Gayat E, Poss J, Schaubroeck H, Billia F, Marshall JC, Lawler PR. Distinct host-response signatures in circulatory shock: a narrative review. Intensive Care Med Exp. 2023 Aug 18;11(1):50. doi: 10.1186/s40635-023-00531-5. PMID 37592121
- [Background] Sarma D, Jentzer JC, Soussi S. Cardiogenic shock: a major challenge for the clinical trialist. Curr Opin Crit Care. 2023 Aug 1;29(4):371-380. doi: 10.1097/MCC.0000000000001066. Epub 2023 Jun 19. PMID 37338937
- [Background] Mebazaa A, Soussi S. Precision Medicine in Cardiogenic Shock: We Are Almost There! JACC Heart Fail. 2023 Oct;11(10):1316-1319. doi: 10.1016/j.jchf.2023.06.024. Epub 2023 Aug 16. No abstract available. PMID 37589609
- [Background] Soussi S, Collins GS, Juni P, Mebazaa A, Gayat E, Le Manach Y. Evaluation of Biomarkers in Critical Care and Perioperative Medicine: A Clinician's Overview of Traditional Statistical Methods and Machine Learning Algorithms. Anesthesiology. 2021 Jan 1;134(1):15-25. doi: 10.1097/ALN.0000000000003600. PMID 33216849
- [Derived] Soussi S, Tarvasmaki T, Kimmoun A, Ahmadiankalati M, Azibani F, Dos Santos CC, Duarte K, Gayat E, Jentzer JC, Harjola VP, Hibbert B, Jung C, Johan L, Levy B, Lu Z, Lawler PR, Marshall JC, Poss J, Sadoune M, Nguyen A, Raynor A, Peoc'h K, Thiele H, Mathew R, Mebazaa A. Identifying biomarker-driven subphenotypes of cardiogenic shock: analysis of prospective cohorts and randomized controlled trials. EClinicalMedicine. 2024 Dec 18;79:103013. doi: 10.1016/j.eclinm.2024.103013. eCollection 2025 Jan. PMID 39802301